CLINICAL TRIAL: NCT02741674
Title: National Patient-Centered Clinical Research Network (PCORnet) Bariatric Study
Brief Title: Comparing the Benefits and Harms of Three Types of Weight Loss Surgery -- The PCORnet® Bariatric Study
Acronym: PBS
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Patient-Centered Clinical Research Network (Other); Chicago Area Patient-Centered Outcomes Research Network (CAPriCORN) (Other); Greater Plains Collaborative Clinical Data Research Network (Other); Research Action for Health Network (REACHnet) (Other); Mid-South Clinical Data Research Network (Other); PEDSnet: A Pediatric Learning Health System CDRN (Unknown); New York City Clinical Data Research Network (Other); OneFlorida Clinical Research Consortium (Other); The Patient-Oriented Scalable National Network for Effectiveness Research (Other); PaTH: Towards a Learning Health System Clinical Data Research Network (Unknown); Scalable Collaborative Infrastructure for a Learning Healthcare System (SCILHS) (Unknown); COPD Patient-Powered Research Network (Unknown); Obesity Action Coalition (Unknown); Harvard Pilgrim Health Care (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-1505-30683
Record Dates: First submitted 2016-04-11; First posted 2016-04-18 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Bariatrics; Body Weight; Diabetes Mellitus; Weight Loss; Roux-en-Y Gastric Bypass; Gastric Bypass
Keywords: Observational Study; Comparative Effectiveness Research
MeSH Terms: conditions — Obesity; Body Weight; Diabetes Mellitus; Weight Loss | interventions — Gastric Bypass; Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Roux-en-y gastric bypass (RYGB): 1. Adults and children ages 12 ≤79 years at time of surgery
  2. Had a primary (not revision) Roux-en-y gastric bypass from years 2005-2015 (based on ICD-9-CM, CPT-4, and HCPCS codes)
  3. Have a Body Mass Index (BMI) measurement in the year prior to surgery that is ≥35 kg/m2 for adults and adolescents
  Interventions: Procedure: Roux-en-y gastric bypass (RYGB) - historical
- Adjustable gastric banding (AGB): 1. Adults and children age 12 ≤79 years at time of surgery
  2. Had a primary (not revision) adjustable gastric banding procedure from years 2005-2015 (based on ICD-9-CM, CPT-4, and HCPCS codes)
  3. Have a Body Mass Index (BMI) measurement in the year prior to surgery that is ≥35 kg/m2 for adults and adolescents
  Interventions: Procedure: Adjustable gastric banding (AGB) - historical
- Sleeve gastrectomy (SG): 1. Adults and children age 12 ≤79 years at time of surgery
  2. Had a primary (not revision) sleeve gastrectomy from years 2005-2015 (based on ICD-9-CM, CPT-4, and HCPCS codes)
  3. Have a Body Mass Index (BMI) measurement in the year prior to surgery that is ≥35 kg/m2 for adults and adolescents
  Interventions: Procedure: Sleeve gastrectomy (SG) - historical

INTERVENTIONS:
Procedure: Roux-en-y gastric bypass (RYGB) - historical — Participant has had RYGB, as identified using existing data
  Groups: Roux-en-y gastric bypass (RYGB)
Procedure: Adjustable gastric banding (AGB) - historical — Participant has had AGB, as identified using existing data
  Groups: Adjustable gastric banding (AGB)
Procedure: Sleeve gastrectomy (SG) - historical — Participant has had SG, as identified using existing data
  Groups: Sleeve gastrectomy (SG)

SUMMARY:
The main goal of this research project is to conduct a comparative effectiveness research study involving existing data in the PCORnet Common Data Model to provide accurate estimates of the 1-, 3-, and 5-year benefits and risks of the three most common bariatric procedures - Roux-en-y gastric bypass, adjustable gastric banding, and sleeve gastrectomy - with a focus on outcomes that are important to adults and adolescents with severe obesity: 1) changes in weight, 2) rates of remission and relapse of diabetes, and 3) major adverse events.

DETAILED DESCRIPTION:
The main aims of this study will compare the effectiveness and safety of the three most common bariatric surgical procedures: Roux-en-y gastric bypass (RYGB), adjustable gastric banding (AGB), and sleeve gastrectomy (SG).

Question (Aim) 1: To what extent does weight loss and weight regain differ across the three bariatric surgical procedures at 1, 3, and 5 years? This aim addresses the primary outcome of interest among most patients seeking bariatric surgery - the differential impact of these procedures on maximum weight loss as well as the extent of longer-term weight regain. We will also explore the heterogeneity in weight loss and regain across several key subgroups that may have differential response to surgical treatment, specifically groups defined by age, race/ethnicity, baseline BMI, smoking status, and pre-operative comorbidities.

Question (Aim) 2: To what extent do these bariatric procedures differ on improvements in diabetes risk at 1, 3, and 5 years? Among patients with diabetes, remission or "cure" of their disease (defined as HbA1c <6.5% off diabetes medications) has been cited as the most important outcome of bariatric surgery. Thus, we will examine the comparative effect of these procedures on rates of diabetes remission as well as relapse (recurrence). Secondary analyses will examine the comparative impact of the procedures on glycemic control independent of diabetes remission.

Question (Aim) 3: What is the frequency of major adverse events following these three different bariatric surgical procedures at 1, 3, and 5 years? We will examine four important adverse event outcome categories across the three procedures: 1) short- and long-term (1, 3, and 5 year) mortality rates, 2) a composite end point of 30-day major adverse outcomes: based on the definition used in the Longitudinal Assessment of Bariatric Surgery (LABS) study that included death; venous thromboembolism; percutaneous, endoscopic, or operative subsequent intervention; and failure to be discharged from the hospital; 3) subsequent hospitalization (any hospitalization following initial surgery); and 4) subsequent reoperation/reintervention: defined as any additional bariatric procedure and other procedures related to device removals, gastric revisions, abdominal or incisional hernia repair, laparoscopy or laparotomy, and percutaneous endoscopic gastrostomy tube placements.

Question (Aim) 4: To what extent do bariatric surgery outcomes explored in Aims 1-3 differ with respect to baseline depression diagnosis at 1, 3, and 5 years after surgery?

Question (Aim) 5: To what extent do bariatric surgery outcomes explored in Aims 1-3 differ with respect to race and ethnicity at 1, 3, and 5 years after surgery?

ELIGIBILITY:
ALL STUDY AIMS

* Inclusion Criteria:

  * Adults and children ages 12 ≤79 years at time of surgery
  * Had a primary (not revision) bariatric procedure from years 2005-2015 of one of three types:

    1. Roux-en-y gastric bypass (RYGB)
    2. Adjustable gastric banding (AGB)
    3. Sleeve gastrectomy (SG)
  * Have a Body Mass Index (BMI) measurement in the year prior to surgery that is ≥35 kg/m2
* Exclusion Criteria:

  * First bariatric procedure during the study period is a revision procedure, a vertical banded gastroplasty procedure or Biliopancreatic Diversion Procedure
  * Have multiple bariatric procedures coded on the same day
  * Have a diagnosis related to GI cancer occurring on day of surgery or during index hospitalization (Diagnosis determined using International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM)
  * Emergency department visit on the same day as hospitalization for bariatric procedure

ADDITIONAL INCLUSION CRITERIA FOR AIM 2 (Diabetes)

• Eligible patients must have uncontrolled or medication-controlled diabetes at the time of surgery.

* Hemoglobin A1c (HbA1c) ≥6.5 % at the most recent measurement prior to surgery, or
* Current prescription for diabetes medication at the time of surgery with the most recent HbA1c <6.5% Patients taking only metformin will be excluded unless they also have an ICD-9-CM code for Diabetes (250.x) or have HbA1c >=6.5% in the year prior to surgery. This includes patients with polycystic ovarian syndrome (PCOS).

ADDITIONAL INCLUSION CRITERIA FOR AIM 3 (Adverse Events)

* Eligible patients must be linked to relevant data sources:

  * State or national death index (mortality outcomes);
  * Payer data/insurance claims (for Adverse Events outcomes)
* Patients must be aged 20 through 79 years of age at time of surgery.

ADDITIONAL EXCLUSION CRITIERA FOR AIM 3 (Adverse Events)

* Exclude any patient with >=365 inpatient hospitalization days in the year prior to surgery.
* Exclude any patient without male or female sex indicated in the study data

AIM 4 (Surgery Outcomes and Baseline Depression) and AIM 5 (Surgery Outcomes and Race/Ethnicity): Inclusion criteria for Aims 1, 2, and 3 will be used for the outcomes from these aims.

ADDITIONAL INCLUSION CRITERIA FOR AIM 5 (Surgery Outcomes and Race/Ethnicity)

• Race and ethnicity available in study data

Ages: 12 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are children and adults (aged 12 through 79 years of age) who have undergone one of the three most common bariatric procedures performed in the United Sates - Roux-en-y gastric bypass, adjustable gastric banding, and sleeve gastrectomy. The population will be identified using participating sites' PCORnet Common Data Model (CDM).
Sampling Method: Non-Probability Sample
Enrollment: 65093 (Actual)
Dates: Start 2016-02; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 1, 3, and 5 years after primary bariatric procedure
  Change in Body Mass Index (BMI)
Diabetes Remission | 1, 3, and 5 years after primary bariatric procedure
  Remission of diabetes after primary bariatric procedure. Defined as individual no longer using any diabetes medication for at least 3 months and hemoglobin A1c (HbA1c) <6.5% after 3 months off of diabetes medication.
Reoperation/Rehospitalization Rate | 1, 3, and 5 years after primary bariatric procedure
  Reoperation: Any additional bariatric procedure and other procedures related to device removals, gastric revisions, abdominal or incisional hernia repair, laparoscopy or laparotomy, and percutaneous endoscopic gastrostomy tube placements.
  Rehospitalization: Any inpatient hospitalization following surgery that is not associated with a delivery, miscarriage, or abortion procedure.

SECONDARY OUTCOMES:
Weight regain | 3 and 5 years after primary bariatric procedure
  At 3 and 5 years after primary bariatric procedure; estimated as percent regain from the maximum weight (in kg) loss in the first 2 years following bariatric surgery.
Diabetes relapse | 1, 3 and 5 years after primary bariatric procedure
  Diabetes relapse defined as restarting diabetes medications or HbA1c >=6.5%
Change in hemoglobin A1C (HbA1c) | 1, 3, and 5 years after primary bariatric procedure
  Change in HbA1c measures.
Mortality Rate | 1, 3, and 5 years after primary bariatric procedure
  Any death during the study period
Composite Adverse Event | 30-days after primary bariatric procedure
  Event is defined using criteria from the Longitudinal Assessment of Bariatric Surgery (LABS) study and includes death; venous thromboembolism; percutaneous, endoscopic, or operative subsequent intervention; and, failure to be discharged from the hospitalization where the bariatric surgery was performed

CONTACTS AND LOCATIONS:
Overall Officials: David E. Arterburn, MD, MPH, Principal Investigator — Kaiser Permanente; Kathleen M. McTigue, MD, MS, MPH, Principal Investigator — University of Pittsburgh; Neely A. Williams, M.Div, Principal Investigator — Mid-South CDRN

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toh S, Rasmussen-Torvik LJ, Harmata EE, Pardee R, Saizan R, Malanga E, Sturtevant JL, Horgan CE, Anau J, Janning CD, Wellman RD, Coley RY, Cook AJ, Courcoulas AP, Coleman KJ, Williams NA, McTigue KM, Arterburn D, McClay J; PCORnet Bariatric Surgery Collaborative. The National Patient-Centered Clinical Research Network (PCORnet) Bariatric Study Cohort: Rationale, Methods, and Baseline Characteristics. JMIR Res Protoc. 2017 Dec 5;6(12):e222. doi: 10.2196/resprot.8323. PMID 29208590
- [Result] McTigue KM, Wellman R, Nauman E, Anau J, Coley RY, Odor A, Tice J, Coleman KJ, Courcoulas A, Pardee RE, Toh S, Janning CD, Williams N, Cook A, Sturtevant JL, Horgan C, Arterburn D; PCORnet Bariatric Study Collaborative. Comparing the 5-Year Diabetes Outcomes of Sleeve Gastrectomy and Gastric Bypass: The National Patient-Centered Clinical Research Network (PCORNet) Bariatric Study. JAMA Surg. 2020 May 1;155(5):e200087. doi: 10.1001/jamasurg.2020.0087. Epub 2020 May 20. PMID 32129809
- [Result] Courcoulas A, Coley RY, Clark JM, McBride CL, Cirelli E, McTigue K, Arterburn D, Coleman KJ, Wellman R, Anau J, Toh S, Janning CD, Cook AJ, Williams N, Sturtevant JL, Horgan C, Tavakkoli A; PCORnet Bariatric Study Collaborative. Interventions and Operations 5 Years After Bariatric Surgery in a Cohort From the US National Patient-Centered Clinical Research Network Bariatric Study. JAMA Surg. 2020 Mar 1;155(3):194-204. doi: 10.1001/jamasurg.2019.5470. PMID 31940024
- [Result] Arterburn D, Wellman R, Emiliano A, Smith SR, Odegaard AO, Murali S, Williams N, Coleman KJ, Courcoulas A, Coley RY, Anau J, Pardee R, Toh S, Janning C, Cook A, Sturtevant J, Horgan C, McTigue KM; PCORnet Bariatric Study Collaborative. Comparative Effectiveness and Safety of Bariatric Procedures for Weight Loss: A PCORnet Cohort Study. Ann Intern Med. 2018 Dec 4;169(11):741-750. doi: 10.7326/M17-2786. Epub 2018 Oct 30. PMID 30383139
- [Result] Inge TH, Coley RY, Bazzano LA, Xanthakos SA, McTigue K, Arterburn D, Williams N, Wellman R, Coleman KJ, Courcoulas A, Desai NK, Anau J, Pardee R, Toh S, Janning C, Cook A, Sturtevant J, Horgan C, Zebrick AJ, Michalsky M; PCORnet Bariatric Study Collaborative. Comparative effectiveness of bariatric procedures among adolescents: the PCORnet bariatric study. Surg Obes Relat Dis. 2018 Sep;14(9):1374-1386. doi: 10.1016/j.soard.2018.04.002. Epub 2018 Apr 17. PMID 29793877
- [Result] Coughlin JW, Nauman E, Wellman R, Coley RY, McTigue KM, Coleman KJ, Jones DB, Lewis KH, Tobin JN, Wee CC, Fitzpatrick SL, Desai JR, Murali S, Morrow EH, Rogers AM, Wood GC, Schlundt DG, Apovian CM, Duke MC, McClay JC, Soans R, Nemr R, Williams N, Courcoulas A, Holmes JH, Anau J, Toh S, Sturtevant JL, Horgan CE, Cook AJ, Arterburn DE; PCORnet Bariatric Study Collaborative. Preoperative Depression Status and 5 Year Metabolic and Bariatric Surgery Outcomes in the PCORnet Bariatric Study Cohort. Ann Surg. 2023 Apr 1;277(4):637-646. doi: 10.1097/SLA.0000000000005364. Epub 2022 Jan 19. PMID 35058404
- [Result] Coleman KJ, Wellman R, Fitzpatrick SL, Conroy MB, Hlavin C, Lewis KH, Coley RY, McTigue KM, Tobin JN, McBride CL, Desai JR, Clark JM, Toh S, Sturtevant JL, Horgan CE, Duke MC, Williams N, Anau J, Horberg MA, Michalsky MP, Cook AJ, Arterburn DE, Apovian CM; PCORnet Bariatric Study Collaborative. Comparative Safety and Effectiveness of Roux-en-Y Gastric Bypass and Sleeve Gastrectomy for Weight Loss and Type 2 Diabetes Across Race and Ethnicity in the PCORnet Bariatric Study Cohort. JAMA Surg. 2022 Oct 1;157(10):897-906. doi: 10.1001/jamasurg.2022.3714. PMID 36044239
- See also: PCORnet Bariatric Surgery Collaborative. The National Patient-Centered Clinical Research Network (PCORnet) Bariatric Study Cohort: Rationale, Methods, and Baseline Characteristics. (Journal link) — http://www.researchprotocols.org/2017/12/e222/
- See also: PCORnet Bariatric Surgery Collaborative. The National Patient-Centered Clinical Research Network (PCORnet) Bariatric Study Cohort: Rationale, Methods, and Baseline Characteristics. (PMC link) — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5736875/
- See also: Comparing the 5-Year Diabetes Outcomes of Sleeve Gastrectomy and Gastric Bypass: The National Patient-Centered Clinical Research Network (PCORNet) Bariatric Study — https://pubmed.ncbi.nlm.nih.gov/32129809/
- See also: Comparative effectiveness of bariatric procedures among adolescents: the PCORnet bariatric study. — https://pubmed.ncbi.nlm.nih.gov/29793877/
- See also: Interventions and Operations 5 Years After Bariatric Surgery in a Cohort From the US National Patient-Centered Clinical Research Network Bariatric Study — https://pubmed.ncbi.nlm.nih.gov/31940024/
- See also: Comparative Effectiveness and Safety of Bariatric Procedures for Weight Loss: A PCORnet Cohort Study — https://pubmed.ncbi.nlm.nih.gov/30383139/
- See also: Preoperative Depression Status and 5 Year Metabolic and Bariatric Surgery Outcomes in the PCORnet Bariatric Study Cohort — https://pubmed.ncbi.nlm.nih.gov/35058404/

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT02741674/SAP_000.pdf